CLINICAL TRIAL: NCT00713349
Title: A Randomized, Evaluator Blinded, Controlled Study of the Effect of Xenaderm® Ointment Vehicle Versus White Petrolatum on Healing of Induced Thermal Wounds
Brief Title: Controlled Study of the Effect of Xenaderm® Ointment Vehicle Versus White Petrolatum on Healing
Status: Completed | Phase: Phase 2 | Type: Interventional
Sponsor: Healthpoint (Industry)
Responsible Party: Sponsor
Allocation: Randomized | Model: Single Group | Masking: Single | Purpose: Treatment
Other Study IDs: 011-101-09-004; NCT00693810 (obsolete NCT alias)
Record Dates: First submitted 2008-07-09; First posted 2008-07-11 (Estimated); Results first posted 2013-12-06 (Estimated); Last update posted 2013-12-06 (Estimated); Status verified 2013-10

CONDITIONS: Wounds
Keywords: White; Petrolatum; Xenaderm; Vehicle; Partial thickness wounds; Healing; Cryo-surgery
MeSH Terms: conditions — Wounds and Injuries | interventions — Granulex

STUDY DESIGN:
Who Masked: Investigator
Oversight: Data Monitoring Committee: No

ARMS (2):
- 1 (Other): Xenaderm Vehicle
  Interventions: Drug: Xenaderm Vehicle
- 2 (Placebo Comparator): Placebo Comparator
  Interventions: Other: Placebo comparator

INTERVENTIONS:
Drug: Xenaderm Vehicle — Ointment to be applied three times a day on cryo-surgery wound for 21 days.
  Other Names: Subject acts as own control
  Arms: 1
Other: Placebo comparator — Ointment to be applied three times a day on cryo-surgery wound for 21 days.
  Other Names: Subject acts as own control
  Arms: 2

SUMMARY:
The objective of the study is to compare the healing of wounds induced by cryo-injury when treated with white petrolatum versus an ointment vehicle.

ELIGIBILITY:
Inclusion Criteria:

Subjects will be considered qualified for enrollment if they:

* Provide written informed consent, which will consist of reading, signing, and dating the informed consent document after the Investigator, sub-Investigator or other designated study staff member has explained the study procedures, risks and contact information.
* Are male or female, ≥ 18 years of age, of any race.
* Are willing to attend all required study visits, and to comply with study procedures.
* Meet none of the exclusion criteria (any single exclusion criterion which is met by a potential subject will disqualify that subject from participation in this study).

Exclusion Criteria:

Subjects will be considered NOT qualified for enrollment if they:

* Have a history of dermatomyositis, systemic sclerosis, scleroderma, Sjögren's syndrome, systemic lupus erythematosis, discoid lupus, Ehler's Danlos disease, icthyosis vulgaris, vasculitis or bleeding disorders (coagulopathies).
* Have any dermatologic disease which may be aggravated or provoked by the wounding procedure, such as Lichen Planus, Psoriasis or Vitiligo.
* Have Fitzpatrick scale skin type 6 (never sunburns, deeply pigmented).
* Are at risk of keloid or hypertrophic scar formation, based on personal history, family history, or brief skin exam (conducted at the screening visit to look for keloids or hypertrophic scars).
* Have been treated within the last three months for uncontrolled diabetes mellitus, peripheral vascular disease, vitamin C deficiency, connective tissue disorders, or any other disease process that impedes wound healing.
* Are taking concomitant medications at doses which are known to interfere with healing, such as non-steroidal anti-inflammatory drugs, anti-neoplastic drugs, or immunosuppressive drugs.
* Are using topical glycolic acid products, alpha-hydroxy acid products, retinoids or chemical peel agents in the treatment areas.
* Are using systemic steroids or immunosuppressant agents, or have used these drugs within the past three months.

Min Age: 18 Years | Sex: All | Healthy Volunteers: Yes
Age Groups: Adult, Older Adult
Enrollment: 25 (Actual)
Dates: Start 2008-06; Primary Completion 2008-08 (Actual); Study Completion 2008-09 (Actual)

CONTACTS AND LOCATIONS:
Overall Officials: Herbert R Slade, MD, Study Chair — Healthpoint; D. Innes Cargill, PhD, Study Director — Healthpoint; Steven R Feldman, MD, PhD, Principal Investigator — Wake Forest
Locations (1):
- Dept. of Dermatology, Wake Forrest School of Medicine, Winston-Salem, North Carolina, United States

RESULTS

PARTICIPANT FLOW:
Recruitment Details: Healthy adult volunteers, 18 years of age and older
Pre-assignment Details: Each subject acting as their own control
Groups:
- Vehicle vs. Placebo: Xenaderm Vehicle and White Petrolatum as Placebo Comparator
  Xenaderm Vehicle : Ointment to be applied three times a day on cryo-surgery wound for 21 days.
  White Petrolatum : Ointment to be applied three times a day on cryo-surgery wound for 21 days
  Each subject acting as their own control
Period: Overall Study
Arm/Group | Vehicle vs. Placebo
Started | 25
Completed | 24
Not Completed | 1
Not completed — Protocol Violation | 1

BASELINE CHARACTERISTICS:
Arm/Group | Vehicle vs. Placebo
Number analyzed (Participants) | 25
Age, Categorical [Count of Participants; unit: Participants]
  <=18 years | 1
  Between 18 and 65 years | 24
  >=65 years | 0
Age Continuous [Mean (Standard Deviation); unit: years] | 43 (12.1)
Sex: Female, Male [Count of Participants; unit: Participants]
  Female | 22
  Male | 3
Region of Enrollment [Number; unit: participants]
  United States | 25

OUTCOME MEASURES:

1. Primary Outcome: Complete Wound Closure
Description: Each subject acting as their own control
Time Frame: 21 Days
Measure: Mean (Standard Deviation); unit: days
Groups:
- Vehicle: Xenaderm Ointment Vehicle : each subject acting as their own control
- Placebo Control: White Petrolatum : each subject acting as their own control
Arm/Group | Vehicle | Placebo Control
Number analyzed (Participants) | 24 | 24
days | 14.8 (1.1) | 14.9 (1.3)

ADVERSE EVENTS:
Time Frame: 21 days
Arm/Group | Vehicle | Placebo Control
Serious Adverse Events (participants affected / at risk) | 0/25 | 0/25
Other Adverse Events (participants affected / at risk) | 6/25 | 6/25
OTHER ADVERSE EVENTS (reported when occurring in more than 5% of participants in an arm); cells are participants affected of the arm's N at risk (number of events):
Term (organ system) | Vehicle (N=25) | Placebo Control (N=25)
Skin and subcutaneous tissue disorders (Skin and subcutaneous tissue disorders) | 6 (6) | 6 (6) — Most frequently reported adverse events were in the skin and subcutaneous disorders group; most frequently reported were due to reactions to adhesive of the band-aid: erythema, itching, bleeding, burning; all were assessed unrelated to test articles.

CERTAIN AGREEMENTS:
Principal investigators are sponsor employees: No; Agreement restricts PI disclosure of results: Yes; Restriction type: embargo of 60 days or less